CLINICAL TRIAL: NCT00231933
Title: Culturally-responsive, Person-centered Care for Psychosis
Brief Title: Culturally Responsive Person-Centered Care for Psychosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0502027488; R01MH067687 (NIH); DSIR 82-SESC
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Psychotic Disorders
Keywords: Person-centered Care; Recovery; Disparities; Culturally Responsive Care; Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Participants will receive standard care incorporating illness management recovery
  Interventions: Behavioral: Illness management recovery (IMR)
- 2 (Experimental): Participants will receive illness management recovery plus person-centered planning
  Interventions: Behavioral: Person-centered planning (PCP); Behavioral: Illness management recovery (IMR)
- 3 (Experimental): Participants will receive illness management recovery plus person-centered planning and community integration
  Interventions: Behavioral: Person-centered planning (PCP); Behavioral: Community integration (CI); Behavioral: Illness management recovery (IMR)

INTERVENTIONS:
Behavioral: Person-centered planning (PCP) — PCP aids participants in discovering a vision of a desirable future and developing a plan for achieving that goal. Techniques include providing direction in the planning process, involving significant others, generating focus on assets and capacities, identifying and providing access to integrated community settings, and promoting acceptance of set backs as part of the path to success.
  Arms: 2; 3
Behavioral: Community integration (CI) — CI includes recovery group sessions and community integration activities.
  Arms: 3
Behavioral: Illness management recovery (IMR) — IMR focuses on nine topic areas: recovery strategies; facts about psychosis; a stress-vulnerability model; building social support; reducing relapses; effective use of medications; coping with stress; coping with problems or symptoms; and meeting health care needs.

SUMMARY:
This study will compare standard individualized care to person-centered care and community-integrating care for treating psychosis in adults of Hispanic or African descent.

DETAILED DESCRIPTION:
Patient-centered care is a type of customized mental health care that is based on each individual's needs, values, and preferences. This type of care has become increasingly important, especially for members of ethnic minorities. However, although this type of care is, in theory, more effective than standard, less personalized care in treating psychotic disorders, there is a significant gap between theory and practice. Research has shown that this gap is particularly evident in the treatment of psychotic disorders in individuals of ethnic backgrounds. This study will address these disparities by comparing the effectiveness of standard individualized care versus person-centered care and community-integrating care in treating psychosis in adults of Hispanic and African descents.

This open-label study will consist of two phases. In Phase I, interview data on self-management of mental illness and treatment seeking behaviors will be collected and analyzed. In Phase II, participants from two urban mental health centers will be randomly assigned to receive one of three treatment combinations: standard care incorporating illness management recovery (IMR); IMR plus person-centered planning (PCP); or IMR plus PCP and community integration (CI). IMR will focus on nine topic areas: recovery strategies; facts about psychosis; a stress-vulnerability model; building social support; reducing relapses; effective use of medications; coping with stress; coping with problems or symptoms; and meeting health care needs. PCP will aid participants in discovering a vision of a desirable future and developing a plan for achieving that goal. Techniques will include providing direction in the planning process, involving significant others, generating focus on assets and capacities, identifying and providing access to integrated community settings, and promoting acceptance of setbacks as part of the path to success. CI will include recovery group sessions and community integration activities. Recovery groups will consist of 10 to 12 people per group, and will aid participants in asserting the skills they learned in IMR and PCP. Community integration activities will entail a variety of excursions and social and recreational activities in the community to promote community involvement and acquisition of social roles. All treatments will last a total of 6 months. Assessments of psychiatric symptoms, social functioning, quality of life, and community integration will occur at Month 6 and at a follow-up visit at Month 18.

ELIGIBILITY:
Inclusion Criteria:

* Of Hispanic and/or African origin
* DSM-IV diagnosis of an axis I psychotic disorder (e.g., schizophrenia, schizoaffective disorder, or bipolar disorder with psychotic features)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2005-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Psychiatric symptoms | Measured at Months 6 and 18
Social functioning | Measured at Months 6 and 18
Quality of life | Measured at Months 6 and 18
Community integration | Measured at Months 6 and 18

SECONDARY OUTCOMES:
Collaborative nature of care | Measured at Months 6 and 18
Culturally responsive nature of care | Measured at Months 6 and 18

CONTACTS AND LOCATIONS:
Overall Officials: Larry Davidson, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States